CLINICAL TRIAL: NCT02286141
Title: Evaluation of a Patient-Centered Risk Stratification Method for Improving Primary Care for Back Pain
Brief Title: Matching Appropriate Treatments to Consumers' Healthcare Needs, MATCH
Acronym: MATCH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI NA
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Patients receiving care at primary care clinics randomized to receive the supplemental training on stratified care for back pain through the use of the StartBack Tool will be considered to be a part of the intervention group. Randomization is done at the clinic level and not at the individual patient level.
- Control: Patients receiving care at primary care clinics randomized to receive the standard Group Health training on the updated Guidelines for Back Pain Care will be considered to be a part of the control group. Randomization is done at the clinic level and not at the individual patient level.

SUMMARY:
Back pain is one of the most common, controversial and costly problems in healthcare. Despite numerous studies, care for back pain has deteriorated over time and become much more expensive. The risk stratification approach developed in England and found effective in National Health Service general practices in the UK provides a very promising strategy for improving care for back pain in the U.S.

The MATCH trial will use a cluster randomization design involving 6 primary care clinics at Group Health. Of these 6 clinics, 3 will be randomized to receive Group Health's standard training in the use of Group Health back pain guidelines and 3 clinics will receive this standard training plus supplemental training. Primary care clinicians and physical therapists in the intervention group will receive training in the use of the STarTBack risk stratification strategy for matching the most appropriate evidence-based treatments to the needs of patients in each risk level. We will evaluate the effect of this supplemental training on patient outcomes, clinician and physical therapist knowledge and comfort treating patients with back pain, and utilization of services for back pain.

DETAILED DESCRIPTION:
Many Americans suffer from back pain for which no specific cause has been identified. Doctors in the United States do not have a standard toolkit of helpful treatments for addressing non-specific back pain. This contributes to frustration and unrelieved suffering for many patients and a sense of helplessness for many doctors. Recently, researchers in England developed a tool called "STarT Back" which helps doctors identify the types of treatments that are most likely to help patients with different pain experiences. This tool divides persons with back pain into three categories based on their answers to 9 simple questions about their pain and its effect on their lives. Doctors can then recommend treatments that are most likely to be helpful for patients in each category. This method has not yet been tested in the United States where healthcare is very different than in England. This project will test an enhanced version of the method at Group Health, a healthcare system in Washington State.

OBJECTIVES: A research team at Group Health will test how well an enhanced version of the STarT Back method works for patients with back pain. Since this method is new in the United States it is important to find out if it meets the needs of patients and doctors, and whether it can be easily used in the doctor's office.

The goals of this project are to:

1. Adapt the STarT Back method for use at Group Health, using its computerized health record system.
2. See how well the method works in three Group Health clinics, compared with three similar clinics where the method is not in place. We will learn from patients and doctors whether the method improved the treatment process and provided patients with greater relief from their back pain.
3. Share the results of this study with other groups, including patients, doctors, healthcare leaders, and other scientists.

METHODS: It is important to understand whether using the method helps provide patients with more pain relief and improves their quality of life. We will invite patients visiting their primary care doctors for back pain to take part in the study. We will also ask doctors and care teams from these clinics to be part of this research. Patients who agree to be in the study will be asked questions about their back pain soon after their doctor visit and again 2 and 6 months later. These questions will be asked in a telephone or mailed survey. This information will allow us to see if using this approach in doctors' offices reduces pain and improves quality of life. We will also ask a small number of patients more in-depth questions to find out if there are ways we can improve this approach. Persons with back pain will be part of the research team. They will give their opinions about all details of the study, including the strategy for implementing the approach, the questions we ask patients and doctors, and how we report the results of the study.

ELIGIBILITY:
Inclusion Criteria:

At least one primary care visit at one of the 6 Group Health clinics involved in this study resulting in a clinical Diagnosis of Back Pain.

Exclusion Criteria:

Pregnancy, Blindness, Deafness, Unable to read or speak English, Paralysis, Psychoses, major, Dementia, Severe Vision problems Severe Hearing problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group Health enrollees aged 18 and older who make a visit to one of the six primary care clinics participating in this study that results in a diagnosis of non-specific back pain.
Sampling Method: Non-Probability Sample
Enrollment: 1760 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Back pain related dysfunction | 6 month
  Back-related dysfunction will be measured with the modified Roland Disability Questionnaire ("Roland scale"), which asks whether 23 specific activities were limited due to back pain during the past week (yes or no). This measure has been found to be reliable, valid and sensitive to clinical changes and is appropriate for telephone administration and patients with moderate disability.
Back Pain Symptom Bothersomeness | 6 month
  Symptom bothersomeness will be measured by asking participants to rate how "bothersome" their back pain has been during the previous week on a 0 to 10 scale (0 = "not at all bothersome" and 10 = "extremely bothersome"). This question worked well in our previous trials and is highly correlated with a 0-10 measure of pain intensity (r=0.8 to 0.9). It is also highly correlated with measures of function and other outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Cherkin, PhD, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Hsu C, Evers S, Balderson BH, Sherman KJ, Foster NE, Estlin K, Levine M, Cherkin D. Adaptation and Implementation of the STarT Back Risk Stratification Strategy in a US Health Care Organization: A Process Evaluation. Pain Med. 2019 Jun 1;20(6):1105-1119. doi: 10.1093/pm/pny170. PMID 30272177
- [Derived] Cherkin D, Balderson B, Wellman R, Hsu C, Sherman KJ, Evers SC, Hawkes R, Cook A, Levine MD, Piekara D, Rock P, Estlin KT, Brewer G, Jensen M, LaPorte AM, Yeoman J, Sowden G, Hill JC, Foster NE. Effect of Low Back Pain Risk-Stratification Strategy on Patient Outcomes and Care Processes: the MATCH Randomized Trial in Primary Care. J Gen Intern Med. 2018 Aug;33(8):1324-1336. doi: 10.1007/s11606-018-4468-9. Epub 2018 May 22. PMID 29790073
- [Derived] Suri P, Delaney K, Rundell SD, Cherkin DC. Predictive Validity of the STarT Back Tool for Risk of Persistent Disabling Back Pain in a U.S. Primary Care Setting. Arch Phys Med Rehabil. 2018 Aug;99(8):1533-1539.e2. doi: 10.1016/j.apmr.2018.02.016. Epub 2018 Apr 3. PMID 29625095
- [Derived] Cherkin D, Balderson B, Brewer G, Cook A, Estlin KT, Evers SC, Foster NE, Hill JC, Hawkes R, Hsu C, Jensen M, LaPorte AM, Levine MD, Piekara D, Rock P, Sherman K, Sowden G, Wellman R, Yeoman J. Evaluation of a risk-stratification strategy to improve primary care for low back pain: the MATCH cluster randomized trial protocol. BMC Musculoskelet Disord. 2016 Aug 24;17(1):361. doi: 10.1186/s12891-016-1219-0. PMID 27553626